CLINICAL TRIAL: NCT04207242
Title: Social Media Use of Psoriasis Vulgaris Patients: Multicenter, Survey Work
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Melek Aslan Kayıran, Specialist Dermatologist Doctor, Istanbul Medeniyet University
Other Study IDs: IstanbulMU5
Record Dates: First submitted 2019-12-03; First posted 2019-12-20 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Psoriasis Vulgaris is a chronic, recurrent, inflammatory and hyperproliferative skin disease. Joint involvement is common along with skin involvement. However, metabolic diseases, such as cardiovascular diseases can be accompanied by many systemic diseases, chronic and repetitive due to the quality of life and psychological status of patients can affect. For this reason, patients carry out various research on their diseases on social media and follow programs on these issues in other media such as television and radio. However, there is no study on how much patients are interested in these publications, how much they trust them, and how they reach and organize information via social media. The aim of the study will be to clarify how and how patients with Psoriasis Vulgaris use social media to obtain information about the diagnosis and treatment of their disease, the interaction of patient groups with each other, and how often social media is used, especially in which group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Psoriasis vulgaris patients

Exclusion Criteria:

* patients that don't want to answer questions

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: psoriasis vulgaris patients
Sampling Method: Non-Probability Sample
Enrollment: 1520 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Social media use of psoriasis vulgaris patients, a questionnaire will be asked the patients and try to learn how they use social media for getting information about their disease. | July 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Melek Aslan Kayıran, Istanbul, Turkey (Türkiye)